CLINICAL TRIAL: NCT01572051
Title: Project Osteoarthritis: Recovering Quality of Life Through Education
Acronym: PARQVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: P.A.R.Q.V.E.
Record Dates: First submitted 2012-01-23; First posted 2012-04-05 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2013-10

CONDITIONS: Osteoarthritis; Knee Osteoarthritis
Keywords: osteoarthritis; knee osteoarthritis; education
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Group 1A (3month plus phone) (Experimental): This group will attend to two courses with a 3 month interval between them This group will receive phone calls This group will receive printed material This group will be reassessed in 6 months
  Interventions: Behavioral: Educational Course; Behavioral: Phone Calls; Behavioral: Printed Material
- Group 1B (3month no phone) (Experimental): This group will attend to two courses with a 3 month interval between them This group will NOT receive phone calls This group will receive printed material This group will be reassessed in 6 months
  Interventions: Behavioral: Educational Course; Behavioral: Printed Material
- Group 2A (2month plus phone) (Experimental): This group will attend to two courses with a 2 month interval between them This group will receive phone calls This group will receive printed material This group will be reassessed in 6 months
  Interventions: Behavioral: Educational Course; Behavioral: Phone Calls; Behavioral: Printed Material
- Group 2B (2month no phone) (Experimental): This group will attend to two courses with a 2 month interval between them This group will NOT receive phone calls This group will receive printed material This group will be reassessed in 6 months
  Interventions: Behavioral: Educational Course; Behavioral: Printed Material
- Group 3A (1month plus phone) (Experimental): This group will attend to two courses with a 1 month interval between them This group will receive phone calls This group will receive printed material This group will be reassessed in 6 months
  Interventions: Behavioral: Educational Course; Behavioral: Phone Calls; Behavioral: Printed Material
- Group 3B (1month no phone) (Experimental): This group will attend to two courses with a 1 month interval between them This group will NOT receive phone calls This group will receive printed material This group will be reassessed in 6 months
  Interventions: Behavioral: Educational Course; Behavioral: Printed Material
- Group 4A (no course plus phone) (Experimental): This group will NOT attend to any courses This group will receive phone calls This group will receive printed material This group will be reassessed in 6 months
  Interventions: Behavioral: Phone Calls; Behavioral: Printed Material
- Group 4B (no course no phone) (Experimental): This group will NOT attend to any courses This group will NOT receive phone calls This group will only receive printed material This group will be reassessed in 6 months
  Interventions: Behavioral: Printed Material

INTERVENTIONS:
Behavioral: Educational Course — 2 Educational courses
  Arms: Group 1A (3month plus phone); Group 1B (3month no phone); Group 2A (2month plus phone); Group 2B (2month no phone); Group 3A (1month plus phone); Group 3B (1month no phone)
Behavioral: Phone Calls — Phone Calls
  Arms: Group 1A (3month plus phone); Group 2A (2month plus phone); Group 3A (1month plus phone); Group 4A (no course plus phone)
Behavioral: Printed Material — Printed Material

SUMMARY:
Osteoarthritis (OA) has a major impact on mobility, disability and loss of productivity of patients. Patients can become disabled early in life by OA. The Osteoarthritis Research Society International (OARSI) is concerned to publish guidelines with the respective levels of evidence on the various forms of treatment of osteoarthritis of the knee and hip.It is believed that an education program has a positive impact on quality of life of patients with OA. Changing the habits of those patients is imperative for clinical improvement.

The investigators propose the creation of an educational program consisting of various health professionals so that we can educate the patients about OA disease, and their role in treatment. This program will be administered in a single day and reviewed/reinforced after an interval of time. Half the patients will be monitored monthly by phone when questions specific to each health area will be made to participants. This way we will evaluate the strength of the telephone follow-up. The investigators are going to create educational printed an audiovisual materials for patients, so the patients can access the information given in the theoretical course at home. Calculation of cost-effectiveness and presentation of data to the authorities.

DETAILED DESCRIPTION:
INTRODUCTION

Osteoarthritis (OA) has a major impact on mobility, disability and loss of productivity of patients. Patients can become disabled early in life by OA.(1,2,3) Osteoarthritis is primarily a genetic disease but can be triggered by trauma, intra-articular fractures, axis deviations and joint overloading, including overweight / obesity.

Perhaps the most common type of disease is hand OA, as debilitating to the patient as the changes generated by rheumatoid arthritis. On the other hand, among the most debilitating, is knee OA, that greatly diminish the quality of life of the affected patients. (4) At the Knee Surgery Group of Instituto de Ortopedia e Traumatologia do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (IOT-HCFMUSP) - Orthopedics and Trauma Institute of University of São Paulo's General Hospital - there is a large number of young adult patients who were economically active, until the advent of a joint trauma, which led to early OA. There is also a large number of people seeking our group for a Total Knee Arthroplasty (TKA) without been offered all non-surgical alternatives of treatment. As there are also patients who underwent surgical treatment but suffer from consequences of OA and clinical treatment is their current need. These patients do not receive an appropriate OA clinical care.

Those patients should be reabsorbed by the basic health network. But the patient is returned by the social services at IOT-HCFMUSP, because there is no such reference in the Unified Health System The OARSI is concerned to publish guidelines with the respective levels of evidence on the various forms of treatment of osteoarthritis of the knee and hip. Those guidelines show the importance of education, phone calls, non-drug methods such as physical therapy, exercise, acupuncture, mind and body therapies, the use of insoles and orthotics, canes, crutches and knee pads, and finally the drugs for pain and to slow the progression of the disease. (5,6) It is believed that an education program has a positive impact on quality of life of patients with OA. In England, the simple delivery of educational material showed no different from a course associated with the delivery of educational material. But in countries like Sweden, primary care is concerned to give courses on OA. In France, teaching about the pathology associated with medical consultation was superior to simple medical consultation to improve patients' symptoms and treatment adherence. (6) No paper on only telephone follow-up was performed, but the addition of patient care by phone, always shows better results than a single intervention. (6) The Osteometabolic Diseases Group of IOT-HCFMUSP, initially focused on the care of osteoporosis and other diseases of bone metabolism such as thalassemia and osteogenesis imperfecta. More recently took over the care and research in the treatment of OA, starting with the knee OA, since it's among the most prevalent and debilitating types of OA.(3)

Obesity and knee OA are the most frequent comorbidities in the elderly in the United States (U.S.). Although not presenting the same level of obesity of U.S. patients, our patients with OA also are overweight, and often have diabetes and hypertension. Changing the habits of those patients is imperative for clinical improvement. Those patients should incorporate healthier eating habits as well as daily physical activity. But to change behavior, it is necessary:

* to perceive the problem as important and serious.
* to perceive that behaviour change is beneficial. Patients are more prone to health information when it is presented in terms of potential gain (11) and when these gains are presented in patients of the same sex and race. (12)

We have a diverse population of patients with level of education ranging from illiterate patients at university level. With this diversity of patients, and a number of patients who can easily reach four digits, and the total lack of possibility of referral of patients to primary or secondary care in the city of São Paulo, we designed a pilot program in three phases:

Phase 1 - Creation of an educational program consisting of various health professionals so that we can educate the patients about OA disease, and their role in treatment. This program will be administered in a single day and reviewed / reinforced after an interval of time. Half the patients will be monitored monthly by phone when questions specific to each health area will be made to participants. This way we will evaluate the strength of the telephone follow-up. We're going to create educational printed an audiovisual materials for patients, so they can access the information given in the theoretical course at home. Calculation of cost-effectiveness and presentation of data to the authorities.

Phase 2 - If we can demonstrate effectiveness in improving the quality of life of patients, we will hold training courses for health professionals from the West Region Project to create a system of reference and cross-reference with the primary and secondary care centers. Patients who have been through the course and demonstrate improved quality of life, will be accompanied closer to their homes in the western region of São Paulo.

Phase 3 - Expansion to all the city of São Paulo and other cities.

In this pilot, we focus exclusively on Phase 1.

The variables that can interfere with patient compliance to the program and, therefore, to the final result, are:

* Length of Interval between interventions (1, 2 or 3 months)
* Phone follow-up or not
* Attending the course or just receiving the educational material

GENERAL OBJECTIVES To assess the improvement of quality of life of patients with osteoarthritis exposed to an education program multi-professional and / or telephone follow-up.

Develop knowledge, experience and indicators that support the expansion of the project to:

West Region Project Municipal Programs, State and National.

Subprojects:

Social Work - improving the quality of life by the introduction of leisure Nutrition - Decrease in body mass index (BMI) by improving the quality and quantity of diet.

Physical Therapy - Improves the autonomy, function and pain for the introduction of daily exercise habits.

Occupational Therapy - Improves autonomy, function and pain by improving the ergonomics and-administration of daily tasks.

Physical Education - Improvement of autonomy, function and pain for the introduction of daily exercise habits.

Psychology - Improving quality of life for the patient and behavior change induced by the intervention.

METHODS

Two hundred and forty patients from the public, healthcare at IOT-HCFMUSP, already identified with OA of the knees

Given the inclusion criteria, patients undergo pre-assessment by the group composed of multi-professional teams of physicians, orthopedic surgeons, nutritionists, psychologists, physiotherapists, occupational therapists, social worker, and physical educators:

Orthopedics - We treat patients according to the OARSI guidelines, offering everything at our disposal for the treatment of OA at IOT-HCFMUSP. Thus, the orthopedic surgeon:

1. - request and evaluate exams, and classify the disease by knees x-rays,
2. - prescribe medications to delay the disease (we work with diacerein in our service), analgesics, muscle relaxants, and Non-Steroidal anti-inflammatory Drugs (NSAIDs), if necessary,
3. - prescribe orthotics (insoles, knee pads, sticks and crutches, braces);
4. - will report to Social Security and Departamento de Transportes (DETRAN) - Transports Department (this, if the social services confirm the need);
5. - Apply evaluation questionnaires SF 36, Visual Analog Pain Scale (VAS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) in the first visit and after six months, will make the referral to physiotherapy and physical activity on the network offered by the government, refers to acupuncture and / or dry needling physiatry in the IOT-FMUSP for cardiac evaluation and clearance for physical activity. Apply the Consent Report to patients.

Each of the professional staff will assess the effects of its intervention in a personalized way through a subproject:

Nutritionist - anthropometric Social Worker - Level of education, autonomy and limited mobility to the hospital.

Psychologist - assess cognitive ability, application of World Health Organization Quality of Life (WHOQOL) Physical Therapist - assess range of motion, pain, strength and quality of life.

Occupational Therapy - range of motion and quality of life. Physical Educator - Evaluate the physical capacity and prescribe appropriate exercise for the patient.

The 240 patients will be randomly assigned to 4 groups of 60. 3 groups will be subjected to 2 interventions, varying the time interval between each intervention: Group 1 to 3 months apart Group 2 - 2 months apart Group 3 - 1-month interval

Group 4 will only receive the printed material.

Patient Flow

Interventions take place on Saturdays at IOT-HCFMUSP, using the classrooms and the dependencies of physiotherapy. We will have a "home simulation" to teach ergonomics in the home. The course will take place between 8:00 and 17:00 hours.

Course Schedule - 30 students per week 7:00 Reception of patients 8:00 Opening 8:10 Orthopedics Class 8:30 Psychology Class 9:30 Interval - Morning Snack 10:00 Theoretical Lecture - Physical Therapy 10:20 Theoretical class - Occupational Therapy 10:40 Practices: Physical Therapy (15 students) and Occupational Therapy (15 students) 12:10 Lunch 13:00 Practices: Physical Therapy (15 students) and Occupational Therapy (15 students 14:30 Nutrition 15:20 Physical Education 15:50 Interval - Afternoon Snack 16:20 Fitness with the Physical Educator 16:30 Social service 17:00 Closure

COURSE CONTENT

1 st Intervention

Education program for 8 hours, with the multidisciplinary team, covered the following:

Psychologist the disease, the role of team and patient in treatment and self-care Nutritionist basics of balancing food Social Worker the importance of leisure experiences and advice about places close to home for recreation and physical activity Physiotherapist Importance of exercise, activities to do at home, experiences Occupational therapy how to deal with daily activities and the limitations caused by OA Physical Educator Differences between physical activity and exercise and the importance for patients with OA Orthopaedist what is the disease can be treated as the daily self-care.

The program will take place on Saturdays at IOT - HCFMUSP, from 8 am to 17 pm

50% of all groups (number of 30 patients in each group 1A, 2A, 3A, and 4A) will receive monthly follow-up by phone. Groups 1B, 2B, 3B, and 4B, will not receive phone calls.

2nd Intervention Education program for 8 hours, with the multidisciplinary team in order to check and reinforce learning of the first intervention.

Psychologist The disease, the role of team and patient in treatment and self-care

Nutritionist Check how patients are feeding anthropometric measures +

Social Worker Check the difficulties encountered by the patient access to physical activity and leisure

Physiotherapist Assessment of range of motion more reinforcement orientation exercises

Occupational therapy Check the difficulties encountered by patients in their daily activities

Orthopaedist Check learning about the disease and self-control

Physical Educator Reinforcing the need for physical activity

The program will take place on Saturdays, the premises of the IOT - HC - FMUSP, from 7 am to 16 pm

AGENDA 2nd. INTERVENTION Schedule Activity

07:00 Reception of patients 08:00 Reviews 09:00 Activity 1 - Orthopaedics 09:20 Activity 2 - Nutrition 10:00 Snack 10:30 Activity 3 - Psychology 11:30 Activity 4 - Physical Therapy 12:30 Lunch 13:30 Activity 5 - Occupational Therapy 14:30 Activity 6 - Social Services 15:30 Assessment Program for Patients and Closure

At the end of 6 months, all groups will return to revaluation with all the teams for reassessment and analysis of the results.

All professionals involved in the program will be paid. The medications used are those provided by the HC complex for patients enrolled with a diagnosis of OA. Any medication that is not in the arsenal of Pharmacy HC for normal service to patients with OA will not be prescribed.

To carry out the interventions on Saturdays (Saturdays 12 in total) will require support services that receive extra payment:

* Secretaries
* Food (snacks morning and afternoon + lunch)
* Computer Support

Estimated Number of sample:

This is a pilot study without a similar estimate for the number of patients. The sample was then left with the number 30 for each subgroup.

Statistical Analysis We will use basic descriptive analysis for sample parameters according to collected data, and Student t test and U Mann-Whitney test to compare pre and post-intervention results.

ELIGIBILITY:
Inclusion Criteria:

* Men and women diagnosed with primary or secondary osteoarthritis of the knees,classified as grades I to IV Kelgreen and Lawrence (KL), ie, any degree of knee osteoarthritis

Exclusion Criteria:

* Patients who have psychiatric or neurological disorders, whose symptoms during the evaluation to the school are related or significantly interfere in the functions of attention, memory, logical reasoning, understanding and interaction with the group in order to undermine the assimilation of the guidelines given

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The benefit of Education in the treatment of knee OA | up to12 months
  To access the results of education on the knee OA outcome

SECONDARY OUTCOMES:
The benefit of phone calls in the treatment of knee OA | 3,6 and 12 months
  To access if we can improve knee OA treatment outcomes with phone calls
Length of interval between interventions | 3,6 and 12 months
  To access what's the optimum interval length between interventions
Which is the best education program - Having classes or only receiving printed material? | 3,6 and 12 months
  Which is the best education program - Having classes or only receiving printed material?

CONTACTS AND LOCATIONS:
Overall Officials: Marcia U Rezende, Phd, Principal Investigator — Hospital das Clínicas da Universidade de São Paulo
Locations (1):
- Instituto de Ortopedia e Traumatologia do Hospital das Clínicas da Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] de Rezende MU, de Farias FES, da Silva CAC, Cernigoy CHA, de Camargo OP. Objective functional results in patients with knee osteoarthritis submitted to a 2-day educational programme: a prospective randomised clinical trial. BMJ Open Sport Exerc Med. 2017 Feb 14;2(1):e000200. doi: 10.1136/bmjsem-2016-000200. eCollection 2016. PMID 28879035